CLINICAL TRIAL: NCT06985693
Title: Medipixel XA-Assisted Percutaneous Coronary Intervention in Coronary Artery Disease: A Prospective Multicenter Study
Brief Title: Medipixel XA-Assisted PCI in Coronary Artery Disease
Acronym: MAP I
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHA University (Other)
Responsible Party: Principal Investigator, Seung-Yul Lee, Associate Professor of Internal Medicine, CHA Bundang Medical Center, CHA University, South Korea, CHA University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHAMC IRB 2025-02-065-001
Record Dates: First submitted 2025-05-15; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Percutaneous Coronary Intervention (PCI); Coronary Arterial Disease (CAD)
Keywords: Artificial Intelligence; Quantitative Coronary Analysis; Medipixel; MPXA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Medipixel XA-Assisted PCI Group (Experimental)
  Interventions: Procedure: Medipixel XA-Assisted Percutaneous Coronary Intervention

INTERVENTIONS:
Procedure: Medipixel XA-Assisted Percutaneous Coronary Intervention — Medipixel XA-Assisted Percutaneous Coronary Intervention (MPXA-PCI) is an AI-assisted coronary intervention procedure utilizing Medipixel XA (MPXA), an artificial intelligence-based quantitative coronary analysis (AI-QCA) software. MPXA analyzes angiographic images in real-time to assist in lesion assessment, optimal balloon and stent selection, and procedural decision-making during percutaneous coronary intervention (PCI).
  In this study, all participants will undergo MPXA-assisted PCI, where the software provides automated vessel segmentation, diameter measurement, and lesion quantification to optimize procedural outcomes. Operators will follow a predefined protocol incorporating MPXA measurements for balloon sizing, stent selection, and post-dilation strategies.
  The study evaluates the safety, feasibility, and clinical impact of MPXA-assisted PCI in real-world coronary artery disease patients.
  Other Names: MPXA-PCI

SUMMARY:
This prospective, multicenter, single-arm, interventional study evaluates the effectiveness and safety of Medipixel XA-Assisted Percutaneous Coronary Intervention (MPXA-PCI) in patients with coronary artery disease (CAD). The study aims to assess procedural success rates and clinical outcomes associated with the novel MPXA-assisted PCI strategy in a real-world clinical setting.

A total of 830 patients with de novo coronary lesions eligible for drug-eluting stent (DES) implantation will be enrolled. All participants will undergo MPXA-assisted lesion assessment to optimize balloon and stent selection. The primary outcome is target vessel failure (TVF) at 12 months, defined as a composite of cardiac death, target vessel-related myocardial infarction, and clinically driven target vessel revascularization. Secondary outcomes include procedural success, angiographic results, and periprocedural complications.

This study will provide evidence regarding the clinical applicability and safety of artificial intelligence-assisted quantitative coronary analysis (AI-QCA) technology for optimizing PCI procedures.

ELIGIBILITY:
Inclusion Criteria:

* Silent ischemia, stable or unstable angina, or myocardial infarction
* De novo coronary lesion eligible for DES implantation
* Lesions analyzable by MPXA

Exclusion Criteria:

* Comorbidity with a life expectancy <12 months
* Intolerant of antithrombotic therapy
* Significant anemia, thrombocytopenia, or leucopenia
* History of major hemorrhage (intracranial, gastrointestinal, and so on)
* Chronic total occlusion lesion
* Left main lesion
* Severe calcification needing rotational atherectomy
* Lesions not analyzable by MPXA

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 830 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Target Vessel Failure (TVF) | 12 months post-procedure
  Target vessel failure (TVF) is a composite of cardiac death, target vessel-related myocardial infarction, and clinically driven target vessel revascularization (TVR).

SECONDARY OUTCOMES:
Minimal Lumen Diameter (MLD) Assessed by MPXA | Immediately post-procedure
  Post-PCI minimal lumen diameter as measured by Medipixel XA.
Residual Stenosis (%) Assessed by MPXA | Immediately post-procedure
  Percentage of remaining stenosis in the treated lesion, as analyzed by MPXA.
MPXA Success Rate | Immediately post-procedure
  Defined as residual stenosis <20% as assessed by Medipixel XA and TIMI 3 flow in the target vessel.
Death | 12 months post-procedure
Myocardial Infarction | 12 months post-procedure
Revascularization | 12 months post-procedure
Stent Thrombosis | 12 months post-procedure
Incidence of Periprocedural Complications | Immediately post-procedure
  Rate of complications such as coronary dissection, perforation, and no-reflow phenomenon.
Rate of Proper Pre-Dilation Balloon Selection | Immediately post-procedure
  Proportion of cases where pre-dilation balloon size was chosen according to MPXA analysis.
Rate of Proper Stent Sizing Selection | Immediately post-procedure
  Proportion of cases where the stent size was selected according to MPXA recommendations.
Frequency of Post-Dilation | Immediately post-procedure
  Number of cases where post-dilation was performed
Rate of Proper Post-Dilation Balloon Selection | Immediately post-procedure
  Proportion of cases where the balloon size adhered to MPXA recommendations.

OTHER OUTCOMES:
Types and Frequency of Additional Interventions Following Intravascular Imaging During PCI | Immediately post-procedure
  This outcome measures the types and frequency of additional interventions performed after intravascular imaging during PCI. Additional interventions may include additional pre-dilation, rotational atherectomy, additional device implantation, additional post-dilation, and other procedures.

CONTACTS AND LOCATIONS:
Locations (6):
- South Korea (6):
  - Chung-Ang University Gwangmyeong Hospital, Gwangmyeong, Gyeonggi-do
  - CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do
  - Keimyung University Dongsan Medical Center, Daegu
  - Chonnam National University Hospital, Gwangju
  - Presbyterian Medical Center, Jeonju
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim Y, Yoon HJ, Suh J, Kang SH, Lim YH, Jang DH, Park JH, Shin ES, Bae JW, Lee JH, Oh JH, Kang DY, Kweon J, Jo MW, Yun SC, Park DW, Kim YH, Park SJ, Park H, Ahn JM; FLASH Trial Investigators. Artificial Intelligence-Based Fully Automated Quantitative Coronary Angiography vs Optical Coherence Tomography-Guided PCI: The FLASH Trial. JACC Cardiovasc Interv. 2025 Jan 27;18(2):187-197. doi: 10.1016/j.jcin.2024.10.025. Epub 2024 Oct 30. PMID 39614852
- [Background] Lee SY, Zhang JJ, Mintz GS, Hong SJ, Ahn CM, Kim JS, Kim BK, Ko YG, Choi D, Jang Y, Kan J, Pan T, Gao X, Ge Z, Chen SL, Hong MK. Procedural Characteristics of Intravascular Ultrasound-Guided Percutaneous Coronary Intervention and Their Clinical Implications. J Am Heart Assoc. 2022 Jul 19;11(14):e025258. doi: 10.1161/JAHA.122.025258. Epub 2022 Jul 15. PMID 35861828
- See also: MPXA Official Website — https://medipixel.io/products/medipixelxa/